CLINICAL TRIAL: NCT02039505
Title: Phase III, Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Intravenous MLN0002 (300 mg) Infusion in Induction and Maintenance Therapy in Japanese Subjects With Moderate or Severe Ulcerative Colitis
Brief Title: Phase III Study of MLN0002 (300 mg) in the Treatment of Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002/CCT-101; U1111-1151-6762 (Other: WHO); JapicCTI-142403 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Ulcerative Colitis
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Induction Phase: Cohort 1, Placebo (Placebo Comparator): Vedolizumab placebo-matching, intravenous (IV) infusion, once at Weeks 0, 2 and 6 in the induction phase.
  Interventions: Drug: Vedolizumab placebo
- Induction Phase: Cohort 1, Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once at Weeks 0, 2, and 6 in the induction phase.
  Interventions: Drug: Vedolizumab
- Induction Phase: Cohort 2, Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once at Weeks 0, 2 and 6 in the induction phase.
  Interventions: Drug: Vedolizumab
- Maintenance Phase: Placebo (Experimental): Vedolizumab placebo-matching, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab in induction phase and achieved clinical response at Week 10 and were randomized to receive placebo in maintenance phase.
  Interventions: Drug: Vedolizumab; Drug: Vedolizumab placebo
- Maintenance Phase: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab in induction phase and achieved clinical response at Week 10 and were randomized to receive vedolizumab in maintenance phase.
  Interventions: Drug: Vedolizumab
- Maintenance Phase: Placebo continuation (Placebo Comparator): Vedolizumab placebo-matching, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab placebo-matching in induction phase and achieved clinical response at Week 10 received placebo in maintenance phase without randomization.
  Interventions: Drug: Vedolizumab placebo
- Open-Label Cohort: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once at Weeks 0, 2 and 6 and then every 8 weeks thereafter up to Week 94 in open-label cohort.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion
  Other Names: MLN0002
  Arms: Induction Phase: Cohort 1, Vedolizumab 300 mg; Induction Phase: Cohort 2, Vedolizumab 300 mg; Maintenance Phase: Placebo; Maintenance Phase: Vedolizumab 300 mg; Open-Label Cohort: Vedolizumab 300 mg
Drug: Vedolizumab placebo — Vedolizumab placebo
  Arms: Induction Phase: Cohort 1, Placebo; Maintenance Phase: Placebo; Maintenance Phase: Placebo continuation

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and pharmacokinetics of the vedolizumab (MLN0002) induction and maintenance therapy in Japanese participants with moderate or severe ulcerative colitis (UC).

DETAILED DESCRIPTION:
This study is a phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to examine the efficacy, safety, and pharmacokinetics of MLN0002 (Vedolizumab) in induction and maintenance therapy in Japanese patients with moderately or severely active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, a participant is capable of understanding and complying with protocol requirements.
2. A participant who is capable of entering the signature and the date on the informed consent by himself/herself or by the participant's legally acceptable representative, if applicable, prior to initiation of study procedures.
3. A participant aged 15 to 80 (inclusive) at the time of signing the informed consent (regardless of sexes).
4. A male participant, who has no sterilization history and whose female partner has child-bearing potential, who agreed with taking proper contraception during the period from the time of signing the informed consent form through 6 months after the last dose of study drug.
5. A female participant with child-bearing potential (having no history of sterilization or whose last menstruation was within 2 years) whose male partner is not receiving contraceptive treatment, and agreed to take proper contraception during the period from the time of signing on the informed consent form through 6 months after the last dose of the study drug.
6. Participants with diagnosis of total or left-sided ulcerative colitis (UC) based on the Revised Diagnostic Criteria for UC issued by "Research Group for Intractable Inflammatory Bowel Disease Designated as Specified Disease" by the Ministry of Health, Labor and Welfare (MHLW) of Japan (2012) at least 6 months before the start of administration of the study drug.
7. A participant with moderately or severely active UC as determined by baseline complete Mayo score of 6 to 12 (inclusive) with an endoscopic subscore of ≥2.
8. Participants whose complication of colon cancer or dysplasia had to be ruled out by total colonoscopy at the start of the study drug administration (or the results from total colonoscopy performed within 1 year before giving consent are available), if participants met any of the following criteria; participants with ≥8-year history of total or left-sided colitis, participants aged ≥50 years, or participants with a first-degree family history of colon cancer.
9. Participants meeting the following treatment failure criteria with at least one of the following agents within 5 years before signing on the informed consent:

   1. Corticosteroids

      * Resistance: Participants whose response was inadequate after treatment of ≥40 mg/day for ≥1 week (oral or IV) or 30 to 40 mg/day for ≥2 weeks (oral or IV).
      * Dependence: Participants for which it is difficult to reduce the dosage to <10 mg/day due to recurrence during gradual dose reduction (oral or IV).
      * Intolerance: Participants who were unable to receive continuous treatment due to adverse reactions (e.g., Cushing's syndrome, osteopenia/osteoporosis, hyperglycaemia, insomnia, infection).
   2. Immunomodulators (azathioprine [AZA] or 6- mercaptopurine [6-MP])

      * Refractory: Participants whose response was inadequate after treatment for ≥12 weeks.
      * Intolerance: Participants who were unable to receive continuous treatment due to adverse reactions (e.g., nausea/vomiting, abdominal pain, pancreatitis, liver function test abnormalities, lymphopenia, thiopurine S-methyltransferase genetic mutation, infection).
   3. Tumor necrosis factor-alpha (TNFα) antagonist

      * Inadequate response: Participants whose response was inadequate after the induction therapy in the dosage described in the package insert.
      * Loss of response: Participants who had recurrence during the scheduled maintenance therapy after achievement of clinical response (those who withdrew for other reasons than relapse are not applicable here).
      * Intolerance: Participants who were unable to receive continuous treatment due to adverse reactions (eg, infusion-related reaction, demyelination, congestive heart failure, infection).

Exclusion Criteria:

1. Participants whose partial Mayo score decrease by 3 points or more between screening and the start of study drug administration.
2. Participants having or suspected to have abdominal abscess or toxic megacolon.
3. Participants with a history of subtotal or total colectomy.
4. Participants with ileostomy, colostomy, fistula or severe intestinal stenosis.
5. Participants having a treatment history with natalizumab, efalizumab or rituximab.
6. Participants who started oral 5-ASA, probiotics, or oral corticosteroids (≤30 mg/day) within 13 days before the first dose of the study drug. Participants who have used these drugs for at least 14 days before the first dose of the study drug, and who changed dosage of or discontinued these drugs within 13 days before the first dose of the study drug.
7. Participants who have received 5-ASA, corticosteroid enemas/suppositories, corticosteroid IV infusion, oral corticosteroid at >30 mg/day, drugs for diarrhea-predominant irritable bowel syndrome, or Chinese herbal medicine for the UC treatment (eg, Daikenchuto) within 13 days before the first dose of the study drug.
8. Participants who have used an antidiarrheal drug for 4 or more consecutive days within 13 days before the first dose of the study drug or within 7 days before the first dose of the study drug.
9. Participants who have received AZA or 6-MP within 27 days before the first dose of the study drug However, this will not apply to participants who have used these drugs for 83 or more days before the first dose of the study drug and continued the steady dose administration of the drugs for 27 or more days before the first dose of the study drug.
10. Participants who have received cyclosporine, tacrolimus, methotrexate, tofacitinib or any study drugs of low-molecular compound for UC treatment within 27 days before the first dose of the study drug.
11. Participants who have received adalimumab within 27 days before the first dose of the study drug or any biologic agents other than adalimumab within 55 days before the first dose of the study drug. However, this will not apply to participants who have topically received these drugs (eg., intraocular injection for treatment of age-related macular degeneration).
12. Participants who have received any live-vaccinations within 27 days before the first dose of the study drug.
13. Participants who underwent the enterectomy within 27 days before the first dose of the study drug or those anticipated to require an enterectomy during the study.
14. Participants who have received leukocytapheresis or granulocyte apheresis within 27 days before the first dose of the study drug.
15. Participants who have been infected with an intestinal pathogen including clostridium difficile or cytomegalovirus within 27 days before the first dose of the study drug.
16. Participants with evidence of adenomatous colonic polyps that need to be removed at the start of study drug administration.
17. Participants with a history or a complication of colonic mucosal dysplasia.
18. Participants suspected to have enteritis other than UC.
19. Participants indicated in the screening test as hepatitis B surface (HBs) antigen-positive or hepatitis C virus (HCV) antibody-positive. Participants indicated as hepatitis B core (HBc) antibody-positive or HBs antibody positive even though HBs antigen-negative However, the criteria will not apply to those with only HBs antibody-positive due to hepatitis B virus (HBV) vaccination, HBV-DNA-negative, HCV antigen-negative or HCV-RNA-negative.
20. Participants who have or are suspected to have a history of tuberculosis (including those whose findings in the chest imaging procedure at screening showing anamnesis of tuberculosis). However, the criteria will not apply to those who had completed prophylactic treatment with isoniazid, and who have been receiving prophylactic isoniazid for 21 days or longer before the first dose of the study drug (the latter may initiate study drug administration with screening phase extended to 28 days at maximum for prophylactic treatment to become 21 days or more).
21. Participants indicated as positive in T-SPOT or QuantiFERON at screening test.
22. Participants who have a history or complication of identified congenital or acquired immunodeficiency syndrome (eg, not-classifiable immunodeficiency, human immunodeficiency virus [HIV] infection or organ transplantation).
23. Participants who were affected by extra-intestinal infection (eg, pneumonia, sepsis, active hepatitis or pyelonephritis) within 27 days before the first dose of the study drug.
24. Participants who have treatment history with MLN0002.
25. Nursing mothers during the screening phase, or female participants indicated positive in urine pregnancy test either at the screening or baseline.
26. Participants having serious complications in the heart, lung, liver, kidney, metabolism, gastrointestinal system, urinary system, endocrine system or blood.
27. Participants with a history of an operation requiring general anesthesia within 27 days before the first dose of the study drug, or with a schedule of an operation requiring hospitalization during the study period.
28. Participants having a complication or a history of malignancy However, it will not apply to the following participants;

    * Participants who had a curative resection of localized skin basal cell carcinoma or had completed curative radiotherapy.
    * Participants who have not experienced recurrence for 1 year or longer since completion of curative resection or curative radiotherapy for skin squamous cell carcinoma.
    * Participants who have not experienced recurrence for 3 year or longer since completion of curative resection or curative radiotherapy for intraepithelial carcinoma of uterine cervix.

    For participants having a substantially distant history of malignancy (eg, 10 years or longer without recurrence since treatment completion), the Investigator and the sponsor will discuss to decide eligibility on the basis of type of malignancy and treatment applied.
29. Participants having a history or a complication of the central nervous disorder, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
30. Participants for which any subjective symptoms in the Subjective PML checklist were found at the screening or baseline.
31. Participants for which any of the following laboratory abnormalities were found at the screening;

    * Hemoglobin ≤8 g/dL
    * White blood cells ≤3,000/μL
    * Lymphocytes ≤500/μL
    * Platelets ≤100,000/μL, or ≥1,200,000/μL
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3×upper limit of normal (ULN)
    * Alkaline phosphatase (ALP) ≥3×ULN
    * Creatinine ≥2×ULN
32. Participants having a history or a complication of alcohol dependence or illicit drug use within one year before the first dose of the study drug.
33. Participants having a history or a complication of psychotic disorder that may obstruct compliance with the study procedures.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (59):
- Japan (59):
  - Kasugai-shi, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyota-shi, Aichi-ken
  - Hirosaki-shi, Aomori
  - Sakura-shi, Chiba
  - Matsuyama, Ehime
  - Fukui-shi, Fukui
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Kurume-shi, Fukuoka
  - Fukuyama-shi, Hiroshima
  - Hatsukaichi-shi, Hiroshima
  - Hiroshima, Hiroshima
  - Asahikawa-shi, Hokkaido
  - Hakodate-shi, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai-shi, Hokkaido
  - Akashi-shi, Hyōgo
  - Himeji-shi, Hyōgo
  - Itami-shi, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Komatsu-shi, Ishikawa-ken
  - Marukame-shi, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Fujisawa-shi, Kanagawa
  - Kamakura-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagasaki, Nagasaki
  - Beppu-shi, Ohita
  - Ōita, Ohita
  - Okayama, Okayama-ken
  - Moriguchi-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Suita-shi, Osaka
  - Saga, Saga-ken
  - Tokorozawa-shi, Saitama
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Shimotsuke-shi, Tochigi
  - Adachi-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Edogawa City, Tokyo
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Wakayama, Wakayama
  - Shunan-shi, Yamaguchi
  - Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Naganuma M, Watanabe K, Motoya S, Ogata H, Matsui T, Suzuki Y, Ursos L, Sakamoto S, Shikamura M, Hori T, Fernandez J, Watanabe M, Hibi T, Kanai T. Potential benefits of immunomodulator use with vedolizumab for maintenance of remission in ulcerative colitis. J Gastroenterol Hepatol. 2022 Jan;37(1):81-88. doi: 10.1111/jgh.15667. Epub 2021 Sep 7. PMID 34409654
- [Derived] Nagahori M, Watanabe K, Motoya S, Ogata H, Kanai T, Matsui T, Suzuki Y, Pinton P, Ursos L, Sakamoto S, Shikamura M, Hori T, Fernandez J, Hibi T, Watanabe M. Week 2 Symptomatic Response with Vedolizumab as a Predictive Factor in Japanese Anti-TNFalpha-Naive Patients with Ulcerative Colitis: A post hoc Analysis of a Randomized, Placebo-Controlled Phase 3 Trial. Digestion. 2021;102(5):742-752. doi: 10.1159/000512235. Epub 2021 Jan 15. PMID 33454706
- [Derived] Okamoto H, Dirks NL, Rosario M, Hori T, Hibi T. Population pharmacokinetics of vedolizumab in Asian and non-Asian patients with ulcerative colitis and Crohn's disease. Intest Res. 2021 Jan;19(1):95-105. doi: 10.5217/ir.2019.09167. Epub 2020 Jul 10. PMID 32635680
- [Derived] Motoya S, Watanabe K, Ogata H, Kanai T, Matsui T, Suzuki Y, Shikamura M, Sugiura K, Oda K, Hori T, Araki T, Watanabe M, Hibi T. Vedolizumab in Japanese patients with ulcerative colitis: A Phase 3, randomized, double-blind, placebo-controlled study. PLoS One. 2019 Feb 26;14(2):e0212989. doi: 10.1371/journal.pone.0212989. eCollection 2019. PMID 30807613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 86 investigative sites in Japan from 04 February 2014 to 28 June 2018.
Pre-assignment Details: Participants with moderate to severe ulcerative colitis (UC) were enrolled. 292 participants enrolled in induction phase, 109 participants entered maintenance phase and 259 participants entered open-label cohort and received placebo or vedolizumab 300 mg. Open-label cohort occurred between Week 10 and Week 154 through study with maximum 94 weeks.
Period: Induction Phase (Week 0 to Week 14)
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Started | 82 | 164 | 46 | 0 | 0 | 0 | 0
Completed | 78 | 155 | 36 | 0 | 0 | 0 | 0
Not Completed | 4 | 9 | 10 | 0 | 0 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 2 | 8 | 7 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Major Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Phase (Week 14 to Week 60)
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Started (Participants who achieved clinical response at Week 10 entered into the maintenance phase.) | 0 | 0 | 0 | 42 | 41 | 26 | 0
Completed | 0 | 0 | 0 | 18 | 30 | 12 | 0
Not Completed | 0 | 0 | 0 | 24 | 11 | 14 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 13 | 8 | 12 | 0
Not completed — Pretreatment Event/Adverse Event | 0 | 0 | 0 | 6 | 1 | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 3 | 2 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Open-Label (Week 10 up to Week 154)
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Started (33 out of 292 participants from induction/maintenance phase did not enter the open-label cohort.) | 0 | 0 | 0 | 0 | 0 | 0 | 259
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 188
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 71
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 44
Not completed — Pretreatment Event/Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 19
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Major Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who entered in the induction phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Total
Number analyzed (Participants) | 82 | 164 | 46 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (15.97) | 42.3 (14.42) | 42.4 (15.60) | 42.8 (15.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 65 | 20 | 112
  Male | 55 | 99 | 26 | 180
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 82 | 164 | 46 | 292
Weight [Mean (Standard Deviation); unit: kg] | 60.36 (12.411) | 58.58 (11.640) | 57.74 (10.559) | 58.95 (11.699)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight(kg)/[height(m)^2]
  kg/m^2 | 21.76 (3.660) | 21.72 (3.411) | 21.12 (2.714) | 21.64 (3.382)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 44 | 85 | 23 | 152
  Current smoker | 3 | 9 | 5 | 17
  Ex-smoker | 35 | 70 | 18 | 123
Duration of Ulcerative Colitis (UC) [Mean (Standard Deviation); unit: years] — Mean duration between the first diagnosis of ulcerative colitis and the start of the study was reported.
  years | 8.57 (7.973) | 7.23 (6.230) | 9.19 (7.725) | 7.91 (7.022)
Complete Mayo Score [Mean (Standard Deviation); unit: score on a scale] — The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
  score on a scale | 8.1 (1.50) | 8.3 (1.54) | 8.3 (1.66) | 8.3 (1.54)
Disease Localization [Count of Participants; unit: Participants]
  Total Colitis | 51 | 101 | 32 | 184
  Left-sided Colitis | 31 | 63 | 14 | 108
Extraintestinal Manifestations [Count of Participants; unit: Participants]
  Had No Extraintestinal Manifestations | 66 | 111 | 32 | 209
  Had Extraintestinal Manifestations | 16 | 53 | 14 | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinical Response at Week 10 in Induction Phase
Description: Clinical response is defined as a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores (rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment), a global assessment by the physician, and an endoscopic subscore. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 10
Population: Full analysis set (FAS) included participants who were randomized and received at least one dose of the study drug in the induction phase. The FAS in the induction phase does not include participants allocated in the Cohort 2 in the induction phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164
percentage of participants | 32.9 [22.942 to 44.186] | 39.6 [32.093 to 47.557]
Statistical Analysis 1: Comparison: Induction Phase: Cohort 1, Placebo vs Induction Phase: Cohort 1, Vedolizumab 300 mg; Test type: Superiority; p = 0.2722, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 1.37, 95% CI 2-sided [0.779 to 2.399] — Cochran-Mantel-Haenszel (CMH) test was used for analysis. Prior tumor necrosis factor alpha (TNFα) antagonist use (yes/no) was used as stratification factor

2. Primary Outcome: Percentage of Participants With Clinical Remission at Week 60 in Maintenance Phase
Description: Clinical Remission is defined as a complete Mayo score of ≤2 points and no individual subscore >1 point. Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 60
Population: FAS included participants who were randomized and received at least one dose of the study drug in the maintenance phase. The FAS in the maintenance phase does not include participants who received placebo in the induction phase and were enrolled into the maintenance phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
percentage of participants | 31.0 [17.622 to 47.086] | 56.1 [39.750 to 71.531]
Statistical Analysis 1: Comparison: Maintenance Phase: Placebo vs Maintenance Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.0210, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 2.88, 95% CI 2-sided [1.168 to 7.108] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

3. Primary Outcome: Number of Participants Who Experienced at Least One or More Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From Baseline to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: Safety analysis set included participants who received at least one dose of the study drug in either the induction phase, the maintenance phase or the open-label cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164 | 46 | 42 | 41 | 26 | 259
Participants | 43 | 82 | 33 | 33 | 36 | 18 | 241

4. Primary Outcome: Number of Participants With TEAE Related to Body Weight
Time Frame: From Baseline to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164 | 46 | 42 | 41 | 26 | 259
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAE Related to Vital Signs
Description: Vital signs included body temperature (axilla), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm).
Time Frame: From Baseline to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164 | 46 | 42 | 41 | 26 | 259
Participants | 2 | 5 | 3 | 2 | 2 | 0 | 24

6. Primary Outcome: Number of Participants With TEAE Related to Electrocardiogram (ECG)
Time Frame: From Baseline to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164 | 46 | 42 | 41 | 26 | 259
Participants | 1 | 1 | 0 | 0 | 0 | 1 | 1

7. Primary Outcome: Number of Participants With Markedly Abnormal Laboratory Parameters Values
Description: The laboratory values outside the range (Hemoglobin <=7 g/dL, Lymphocytes <500 /µL, WBC <2000 /µL, Platelets <7.5 10^4/µL, Neutrophils <1000 /µL, alanine aminotransferase (ALT) >3.0 U/L x upper limit of normal (ULN), aspartate aminotransferase (AST) >3.0 U/L x ULN, Total Bilirubin >2.0 mg/dL x ULN, Amylase >2.0 (U/L) x ULN were considered markedly abnormal. Only laboratory parameters with events were represented.
Time Frame: From Baseline to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164 | 46 | 42 | 41 | 26 | 259
Participants
  Hemoglobin (g/dL) <=7 | 1 | 4 | 1 | 0 | 0 | 0 | 6
  Lymphocytes (/µL) <500 | 6 | 2 | 2 | 1 | 0 | 1 | 20
  White Blood Cell (WBC) (/µL) <2000 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils (/µL) <1000 | 1 | 1 | 1 | 1 | 0 | 0 | 4
  Alanine Aminotransferase (ALT) (U/L) >3.0 x ULN | 1 | 0 | 0 | 1 | 0 | 0 | 4
  Aspartate Aminotransferase (AST) (U/L) >3.0 x ULN | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Total Bilirubin (mg/dL) >2.0 x ULN | 0 | 2 | 0 | 0 | 0 | 0 | 1
  Amylase (U/L) >2.0 x ULN | 1 | 2 | 1 | 0 | 0 | 0 | 4

8. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 10 in Induction Phase
Description: as for outcome 2
Time Frame: Week 10
Population: FAS included participants who were randomized and received at least one dose of the study drug in the induction phase. The FAS in the induction phase does not include participants allocated in the Cohort 2 in the induction phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164
percentage of participants | 12.2 [6.006 to 21.286] | 18.3 [12.695 to 25.072]
Statistical Analysis 1: Comparison: Induction Phase: Cohort 1, Placebo vs Induction Phase: Cohort 1, Vedolizumab 300 mg; Test type: Superiority; p = 0.1980, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 1.66, 95% CI 2-sided [0.762 to 3.596] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

9. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 10 in Induction Phase
Description: Mucosal healing is defined as a Mayo endoscopic subscore of ≤1 point. Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Endoscopic findings were scored on a scale from 0 to 3 as follows: 0=Normal or inactive disease; 1=Mild disease (erythema, decreased vascular pattern, mild friability); 2=Moderate disease (marked erythema, lack of vascular pattern, friability, erosions); 3=Severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 10
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg
Number analyzed (Participants) | 82 | 164
percentage of participants | 30.5 [20.796 to 41.638] | 36.6 [29.213 to 44.452]
Statistical Analysis 1: Comparison: Induction Phase: Cohort 1, Placebo vs Induction Phase: Cohort 1, Vedolizumab 300 mg; Test type: Superiority; p = 0.3168, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 1.33, 95% CI 2-sided [0.755 to 2.356] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

10. Secondary Outcome: Percentage of Participants With Durable Clinical Response in Maintenance Phase
Description: Durable clinical response is defined as reduction in complete Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at both Weeks 10 and 60. Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Weeks 10 and 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
percentage of participants | 35.7 [21.551 to 51.974] | 65.9 [49.405 to 79.917]
Statistical Analysis 1: Comparison: Maintenance Phase: Placebo vs Maintenance Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.0067, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 3.48, 95% CI 2-sided [1.407 to 8.626] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

11. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 60 in Maintenance Phase
Description: as for outcome 9
Time Frame: Week 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
percentage of participants | 33.3 [19.567 to 49.549] | 63.4 [46.936 to 77.877]
Statistical Analysis 1: Comparison: Maintenance Phase: Placebo vs Maintenance Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.0066, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 3.49, 95% CI 2-sided [1.409 to 8.642] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

12. Secondary Outcome: Percentage of Participants With Durable Remission in Maintenance Phase
Description: Durable clinical remission is defined as complete Mayo score of ≤2 points and no individual subscore >1 point at both Weeks 10 and 60. Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Weeks 10 and 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
percentage of participants | 16.7 [6.974 to 31.364] | 26.8 [14.221 to 42.944]
Statistical Analysis 1: Comparison: Maintenance Phase: Placebo vs Maintenance Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.2090, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 2.02, 95% CI 2-sided [0.677 to 6.033] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

13. Secondary Outcome: Percentage of Participants With Corticosteroid-Free Remission at Week 60 in Maintenance Phase
Description: Clinical Remission is defined as a complete Mayo score of ≤2 points and no individual subscore >1 point. Corticosteroid-free clinical remission is defined as participants using oral corticosteroids at baseline (Week 0) who discontinued corticosteroids and were in clinical remission at Week 60. Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 60
Population: Participants from FAS included participants who were randomized and received at least one dose of the study drug in the maintenance phase and administered oral corticosteroids concomitantly at Week 0, were analyzed at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 15 | 13
percentage of participants | 20.0 [4.331 to 48.089] | 46.2 [19.223 to 74.865]
Statistical Analysis 1: Comparison: Maintenance Phase: Placebo vs Maintenance Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.1571, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 3.38, 95% CI 2-sided [0.636 to 17.981] — CMH test was used for analysis. Prior TNFα antagonist use (yes/no) was used as stratification factor

14. Secondary Outcome: Serum Vedolizumab Concentration in Induction Phase
Time Frame: Pre-dose at Weeks 2, 6, 10 and 14
Population: Participants from FAS, who received at least one dose of study drug in induction phase for whom sample was available for pharmacokinetic (PK) analysis. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg
Number analyzed (Participants) | 164 | 46
μg/mL
  Week 2: number analyzed (Participants) | 104 | 31
  Week 2 | 31.93 (9.0617) | 33.96 (7.7002)
  Week 6: number analyzed (Participants) | 96 | 28
  Week 6 | 29.58 (12.965) | 31.53 (12.937)
  Week 10: number analyzed (Participants) | 110 | 29
  Week 10 | 31.42 (14.462) | 36.63 (16.058)
  Week 14: number analyzed (Participants) | 45 | 12
  Week 14 | 16.09 (7.3624) | 19.04 (6.6528)

15. Secondary Outcome: Serum Vedolizumab Concentration in Maintenance Phase
Time Frame: Pre-dose at Weeks 2, 6, 10, 14, 22, 30 and 60
Population: Participants from FAS, who were randomized and received at least one dose of the study drug in the maintenance phase for whom sample was available for PK analysis. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
μg/mL
  Week 2: number analyzed (Participants) | 31 | 30
  Week 2 | 32.87 (9.8729) | 34.92 (7.3732)
  Week 6: number analyzed (Participants) | 29 | 27
  Week 6 | 32.80 (12.953) | 35.87 (11.983)
  Week 10: number analyzed (Participants) | 32 | 32
  Week 10 | 39.21 (15.076) | 41.02 (11.955)
  Week 14: number analyzed (Participants) | 27 | 30
  Week 14 | 16.05 (7.4224) | 17.31 (7.1914)
  Week 22: number analyzed (Participants) | 25 | 26
  Week 22 | 2.913 (2.3243) | 14.45 (6.0327)
  Week 30: number analyzed (Participants) | 25 | 25
  Week 30 | 0.2200 (0.48146) | 13.77 (6.3692)
  Week 60: number analyzed (Participants) | 14 | 25
  Week 60 | 0.000 (0.0000) | 21.16 (8.9078)

16. Secondary Outcome: Number of Participants With Anti-vedolizumab Antibodies (AVA) in Induction Phase
Description: Blood samples were collected and tested for serum concentration of anti-vedolizumab antibodies in a laboratory by means of electrochemoluminescent (ECL) assay.
Time Frame: Weeks 0, 10 and 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: Participants who underwent proper AVA test out of "the FAS in the induction phase" and, "the participants who received at least one dose of study drug in the Cohort 2" were analyzed at the given timepoint. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg
Number analyzed (Participants) | 164 | 46
Participants
  Week 0: number analyzed (Participants) | 116 | 36
  Week 0 | 0 | 0
  Week 10: number analyzed (Participants) | 116 | 36
  Week 10 | 1 | 0
  16 Weeks After Last Administration: number analyzed (Participants) | 7 | 7
  16 Weeks After Last Administration | 1 | 1

17. Secondary Outcome: Number of Participants With Anti-vedolizumab Antibodies (AVA) in Maintenance Phase
Description: Blood samples were collected and tested for serum concentration of anti-vedolizumab antibodies in a laboratory by means of ECL assay.
Time Frame: Weeks 0, 10, 30, 60 and 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: Participants who underwent proper AVA test out of the FAS, the participants who received at least one dose of study drug in the maintenance phase were analyzed at the given timepoint. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
Participants
  Week 0: number analyzed (Participants) | 32 | 33
  Week 0 | 0 | 0
  Week 10: number analyzed (Participants) | 32 | 33
  Week 10 | 0 | 0
  Week 30: number analyzed (Participants) | 31 | 33
  Week 30 | 4 | 0
  Week 60: number analyzed (Participants) | 17 | 25
  Week 60 | 1 | 0
  16 Weeks After Last Administration: number analyzed (Participants) | 4 | 2
  16 Weeks After Last Administration | 0 | 0

18. Secondary Outcome: Number of Participants With Neutralizing Anti-vedolizumab Antibodies (AVA) in Induction Phase
Description: Blood samples were collected, and serum neutralizing AVA was determined only for the AVA-positive samples in a laboratory by means of ECL assay.
Time Frame: Weeks 0, 10 and 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: Participants who underwent proper AVA test out of "the FAS in the induction phase" and "the participants who received at least one dose of study drug in the Cohort 2" were analyzed at the given timepoint. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg
Number analyzed (Participants) | 164 | 46
Participants
  Week 0: number analyzed (Participants) | 116 | 36
  Week 0 | 0 | 0
  Week 10: number analyzed (Participants) | 116 | 36
  Week 10 | 1 | 0
  16 Weeks After Last Administration: number analyzed (Participants) | 7 | 7
  16 Weeks After Last Administration | 1 | 1

19. Secondary Outcome: Number of Participants With Neutralizing Anti-vedolizumab Antibodies (AVA) in Maintenance Phase
Description: as for outcome 18
Time Frame: Weeks 0, 10, 30, 60 and 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 42 | 41
Participants
  Week 0: number analyzed (Participants) | 32 | 33
  Week 0 | 0 | 0
  Week 10: number analyzed (Participants) | 32 | 33
  Week 10 | 0 | 0
  Week 30: number analyzed (Participants) | 31 | 32
  Week 30 | 3 | 0
  Week 60: number analyzed (Participants) | 17 | 25
  Week 60 | 0 | 0
  16 Weeks After Last Administration: number analyzed (Participants) | 4 | 2
  16 Weeks After Last Administration | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Induction Phase: Cohort 1, Placebo | Induction Phase: Cohort 1, Vedolizumab 300 mg | Induction Phase: Cohort 2, Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo Continuation | Open-Label Cohort: Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/164 | 0/46 | 0/42 | 0/41 | 0/26 | 0/259
Serious Adverse Events (participants affected / at risk) | 4/82 | 10/164 | 6/46 | 3/42 | 4/41 | 1/26 | 48/259
Other Adverse Events (participants affected / at risk) | 10/82 | 28/164 | 15/46 | 17/42 | 27/41 | 13/26 | 191/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Cohort 1, Placebo (N=82) | Induction Phase: Cohort 1, Vedolizumab 300 mg (N=164) | Induction Phase: Cohort 2, Vedolizumab 300 mg (N=46) | Maintenance Phase: Placebo (N=42) | Maintenance Phase: Vedolizumab 300 mg (N=41) | Maintenance Phase: Placebo Continuation (N=26) | Open-Label Cohort: Vedolizumab 300 mg (N=259)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 6 | 4 | 2 | 2 | 0 | 25
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Granulomatous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuritis cranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Internal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Cohort 1, Placebo (N=82) | Induction Phase: Cohort 1, Vedolizumab 300 mg (N=164) | Induction Phase: Cohort 2, Vedolizumab 300 mg (N=46) | Maintenance Phase: Placebo (N=42) | Maintenance Phase: Vedolizumab 300 mg (N=41) | Maintenance Phase: Placebo Continuation (N=26) | Open-Label Cohort: Vedolizumab 300 mg (N=259)
Viral upper respiratory tract infection (Infections and infestations) | 8 | 23 | 12 | 9 | 18 | 8 | 130
Headache (Nervous system disorders) | 2 | 6 | 3 | 1 | 2 | 2 | 23
Nausea (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 13
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 2 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 18
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 13
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 19
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 14
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 22
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 17
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 16
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2013-11-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02039505/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT02039505/SAP_001.pdf